CLINICAL TRIAL: NCT03996083
Title: A Randomized Controlled Trial to Compare a Multicomponent Exercise Program and a Walking Program in Long-term Nursing Home Residents
Brief Title: Multicomponent Exercise vs Walking Intervention in Nursing Home Residents
Acronym: MCvsW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, Susana Gil, Principal investigator, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2019
Record Dates: First submitted 2019-06-18; First posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Aging
Keywords: aging; nursing homes; accidental falls; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: participants were randomized (in a 1:1 ratio) through sealed opaque envelopes by coin-tossing sequence generation into either the multicomponent or the walking group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent exercise intervention (Experimental): The multicomponent exercise program consisted of strength and balance exercises performed on two non-consecutive days per week and lasting approximately an hour per session. Strength exercises were mainly focused on lower limb strengthening. A gradual and progressive intensity starting at 40% 1-RM and up 70% 1-RM was used. As for balance exercises, the first weeks consisted of mainly less complex static balance exercises and progressed to more complex and dynamic balance exercises. These exercises included standing with their feet together, semi-tandem, tandem and one-legged stand positions and moving on to dynamic exercises (circuits, stepping and so on). Difficulty was increased by reducing arm and base support and by varying the type and complexity of exercises. An individualized progression was applied to each participant based on their progress throughout the intervention.
  Interventions: Other: Multicomponent exercise intervention
- Walking intervention (Experimental): Participants assigned to the walking group walked with the research staff two days per week; additionally, they walked partially supervised by LTNH staff, family members or caregivers the rest of the week. Daily walking goals were set follows: walking between 5 to 10 minutes on the first month, up to 15 minutes on the second, and finally 20 minutes per day on the third month. The final goal was to get as close as possible to the recommendations of engaging in 150 minutes of aerobic exercise per week from the World Health Organization (WHO). Participants were asked to walk as fast as they could and rest was allowed whenever needed. Walking goals were achieved in one or multiple sessions, depending on each participant´s capacities. Those participants that met the walking goals without any rest were encouraged to walk at a faster pace.
  Interventions: Other: Walking intervention

INTERVENTIONS:
Other: Multicomponent exercise intervention — Strength exercises were focused on lower limb strengthening. Individual bilateral intensities were calculated to estimate one repetition maximum (1-RM) for the leg and arm. This test was performed on the 2nd and 7th weeks of the intervention. A gradual and progressive intensity starting at 40% 1-RM and up 70% 1-RM was used. No external loads were applied to the rest of the exercises due to their complex execution technique and subsequent risk of adverse events. In these cases, training progression was achieved through volume (number of repetitions) and execution velocity increments.
  Balance exercises included standing with their feet together, semi-tandem, tandem and one-legged stand positions and moving on to dynamic exercises (circuits, stepping and so on). Difficulty was increased by reducing arm and base support and by varying the type and complexity of exercises. An individualized progression was applied to each participant based on their progress throughout the intervention.
  Arms: Multicomponent exercise intervention
Other: Walking intervention — To comply with the walking goals, walking distance was calculated based on each participant´s performance on the 6-minute walking test and using a rule of thumb. Therefore, every participant had an itinerary to follow to comply with the minimum walking time each week. Distance rather than time was used with participants for practical reasons and the inability of most of them to measure time. Moreover, time and distance were individually adapted according to each participant´s performance on the previous week.
  To ensure that participants complied with the walking goals, each of them (if they were cognitively able) was given a record sheet in which they had to write down their everyday walking routines. In addition, the caregivers were also informed about the walking routines and ensured that those participants who needed close supervision had someone to walk with and filled the sheet of those that were unable to do so.
  Arms: Walking intervention

SUMMARY:
Physical exercise is an important tool to tackle the deleterious effect of aging. However, which is the best exercise intervention is still unknown. Moreover, many exercise interventions are complicated to implement, particularly in nursing homes. In contrast, walking is a simple, natural, and familiar mode of exercise that is well tolerated by older adults. Thus, the objective was to assess and compare the effects of an individualized multicomponent exercise program and an individualized and progressive walking intervention on LTNH residents´ physical and cognitive performance, habitual physical activity, psycho-affective status and quality of life.

DETAILED DESCRIPTION:
The objective was to assess and compare the effects of an individualized multicomponent exercise program and an individualized and progressive walking intervention on LTNH residents´ physical and cognitive performance, habitual physical activity, psycho-affective status and quality of life.

Design: single-blind randomized controlled trial. 81 men and women were randomly assigned to a multicomponent (MG) or a walking (WG) group after baseline measurements. Participants in the MG underwent a twice a week individualised and progressive multicomponent exercise program composed of strength and balance exercises. The walking group was also individualised and walked progressively to up to 20 minutes per day for the 3-month intervention.

The primary outcome was the score on the Short Physical Performance Battery (lower limb strength (time needed to perform five chair stands), static balance (standing with feet together, semi-tandem and tandem positions) and usual gait speed (4m), assessed at baseline and after the intervention. Secondary outcomes included other relevant physical performance tests (Senior Fitness Test, the Berg Balance Scale, handgrip strength, usual gait speed (4m) the instrumented Timed Up and Go test), habitual physical activity (using accelerometers during 7 days), cognitive performance (Montreal Cognitive Assessment test and the Rey Auditory Verbal Learning Test), psycho-affective status (Anxiety and Depression Goldberg Scale, and loneliness using the Jong Gierveld loneliness scale) and quality of life (the Quality of Life Alzheimer´s disease scale). Also frailty and the number of falls and deaths will be registered.

Descriptive statistics were computed and baseline (between group differences) and time effects (within group differences) were checked using Student´s-t test (quantitative variables) or Chi square test (qualitative variables). Intervention effects between groups were assessed by 2-way analysis of variance for repeated measures (group by time interactions). Partial η2 and Cohen´s d was calculated. All the analysis performed under the intention-to-treat principle and significance was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Score ≥ 50 on the Barthel Index (Wade and Collin, 1988)
* ≥ 20 on the MEC-35 test (an adapted version of the Mini Mental State Examination, MMSE, validated in Spanish) (Lobo et al., 1999)
* capable to stand up and walk with or without assistive devices for at least 10 m.

References:

* Wade D.T., Collin C. The Barthel ADL Index: a standard measure of physical disability? Int Disabil Stud. 1988; 10(2):64-7. doi: 10.3109/09638288809164105.
* Lobo A, Saz P, Marcos G, Díaz J.L, de la Camara C, Ventura T, Morales Asín F, Fernando Pascual L, Montañes J.A, Aznar S. Revalidación y normali-zación del Mini-Examen Cognoscitivo (primera versión en castellano del Mini-Mental Status Exa- mination) en la población general geriátrica. Med Clin (Barc). 1999; 112; 767-774

Exclusion Criteria:

* Participants who were clinically unstable or who had any condition in which the medical staff considered it was not in the subject´s best interests to participate were not included in the study.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery | Measurements will be made at baseline and after the intervention (3 months)
  The Short Physical Performance Battery test (SPPB). It assesses Lower extremity function: static balance, gait speed and getting in and out of a chair. The participant undertakes different tests: Side-by-side, semi-tandem and tandem stands (10 seconds); 4 meters walk test at comfortable speed and 5 quickly sit to stand from a chair without upper extremity assistance. The outcome is a score 0-12 points. A higher score means better performance
  Reference:
  Guralnik et al, 1994. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994; 49(2):M85-94. doi: 10.1093/geronj/49.2.M85.

SECONDARY OUTCOMES:
Senior Fitness Test: strength of the upper extremities | Measurements will be made at baseline and after the intervention (3 months)
  Number of arm curls performed in 30 seconds
  Reference:
  Rikli & Jones, 2007. Senior fitness test. Human Kinetics, Champaign; 2001. ISBN 0-7360-3356-4.
Senior Fitness Test: strength of the lower extremities | Measurements will be made at baseline and after the intervention (3 months)
  Number of Chair-stands performed in 30 seconds
  Reference:
  Rikli & Jones, 2007. Senior fitness test. Human Kinetics, Champaign; 2001. ISBN 0-7360-3356-4.
Senior Fitness Test: flexibility | Measurements will be made at baseline and after the intervention (3 months)
  Performed test: chair sit and reach. The participant is sitting and tries to touch the toes. The distance between the fingers and the toes is measured (cm)
  Reference:
  Rikli & Jones, 2007. Senior fitness test. Human Kinetics, Champaign; 2001. ISBN 0-7360-3356-4.
Senior Fitness Test: dynamic balance | Measurements will be made at baseline and after the intervention (3 months)
  8 Foot Up and Go test: The participant from a sitting positions, gets up and walks a 4 foot distance, turns and comes back. Time is measured in seconds.
  Reference:
  Rikli & Jones, 2007. Senior fitness test. Human Kinetics, Champaign; 2001. ISBN 0-7360-3356-4.
Senior Fitness Test: aerobic capacity | Measurements will be made at baseline and after the intervention (3 months)
  Performed test: 6-minutes walking test. The participant walks during 6 minutes as fast as possible without running. The distance is measured in meters
  Reference:
  Rikli & Jones, 2007. Senior fitness test. Human Kinetics, Champaign; 2001. ISBN 0-7360-3356-4.
The Berg Balance Scale | Measurements will be made at baseline and after the intervention (3 months)
  Estimates postural stability using different positions. Construct: Static balance. Scale range (total score): 0-56 (the higher, the better).
  Reference:
  Berg et al, 1992. Measuring balance in the elderly: validation of an instrument. Can J Publ Health. 1992; 83:S7-11
Usual gait speed (4m) | Measurements will be made at baseline and after the intervention (3 months)
  The participants walks at his/her usual and comfortable pace for 4 m, time is measured in seconds.
  Reference:
  Bohannon et al, 1996. Walking speed: reference values and correlates for older adults. J Orthop Sports Phys Ther. 1996; 24(2):86-90. doi: 10.2519/jospt.1996.24.2.86.
The instrumented Timed Up and Go test | Measurements will be made at baseline and after the intervention (3 months)
  The instrumented Timed Up and Go test, using a BTS Biomedical G-WALK triaxial accelerometer and gyroscope, to measure dynamic balance. The participant gets up from a chair, walks 3 meters at a normal pace, turns and walks back to sit down again.
  Reference:
  Mathias et al, 1986. Balance in elderly patients: the "get-up and go" test. Arch Phys Med Rehabil. 1986; 67(6):387-9.
Objectively measured habitual physical activity | Measurements will be made at baseline and after the intervention (3 months)
  Active and sedentary periods during everyday life recorded with an accelerometer (Actigraph GT3X model (Actigraph LLC, Pensacola, FL, USA)) that is worn on the hip with a belt for a 7 day period. The device is set to quantify the number of steps taken per day. In line with that, active-period intensities will be classified following the criteria developed by Freedson et al., 1998 as low, medium or high intensity and measured in minutes.
  Reference:
  Freedson et al, 1988. Calibration of the Computer Science and Applications, Inc. accelerometer. Med Sci Sports Exerc. 1998; 30(5):777-81. doi: 10.1097/00005768-199805000-00021.
Montreal Cognitive Assessment test | Measurements will be made at baseline and after the intervention (3 months)
  It assesses different cognitive domains: attention and concentration, executive functions, memory, language, constructional skills, conceptual thinking, calculations, and orientation. The total possible score is 30 points; a score of 26 or above is considered normal.
  Reference:
  Coen et al, 2016.Strengths and Limitations of the MoCA for Assessing Cognitive Functioning Findings From a Large Representative Sample of Irish Older Adults. Journal of Geriatric Psychiatry and Neurology. 2016; 29(1):18-24. doi: 10.1177/0891988715598236.
Rey Auditory Verbal Learning Test | Measurements will be made at baseline and after the intervention (3 months)
  It measures learning capacity. Evaluates short- and long-term verbal learning assessing the ability to learn a list of 15 common words.
  Reference:
  Lezak MD, Howieson DB, Loring DW. Neuropsychological Assessment. 4th ed. New York: Oxford University Press; 2004
Anxiety and Depression Goldberg Scale | Measurements will be made at baseline and after the intervention (3 months)
  It is used to assess the affective state. This questionnaire includes nine depression and nine anxiety items from the past month.
  Construct: Anxiety and depression.
  Scale range (Subescale score):
  0-9 Anxiety (the higher, the worse). 0-9 Depression (the higher, the worse).
  Reference:
  Goldberg et al, 1988. Detecting anxiety and depression in general medical settings. Br Med J. 1988; 297(6653):897-9. doi:10.1136/bmj.297.6653.897.
Quality of Life Alzheimer´s disease scale | Measurements will be made at baseline and after the intervention (3 months)
  It measures the perceived quality of life, particularly, self-rated quality of life for people with cognitive impairments.
  Construct: Health related quality of life. Scale range (total score): 13-52 (the higher, the better).
  Reference:
  Logsdon et al., 2002. Assessing quality of life in older adults with cognitive impairment. Psychosomatic Medicine. 2002;64:510-519.
de Jong Gierveld loneliness scale | Measurements will be made at baseline and after the intervention (3 months)
  This questionnaire includes characteristics of the social network, background variables, personality characteristics, and evaluative aspects.
  Construct: Loneliness perception. Scale range (total score): 0-11 (the higher, the worse).
  Reference:
  De Jong Gierveld, J. (1987). Developing and testing a model of loneliness. Journal of Personality and Social Psychology, 53(1), 119-128.
Handgrip strength | Measurements will be made at baseline and after the intervention (3 months)
  For that the participant squeezes the dynamometer with maximum isometric effort for about 5 seconds. It measures strength in kg.
  Reference:
  Fess, 1992. Clinical assessment recommendations. 2. Casanova JS, editor. Chicago: American Society of Hand Therapists; 1992. Grip strength; pp. 41-45.
Anthropometric measurements: Height | Measurements will be made at baseline and after the intervention (3 months)
  To measure heigt the participant stands up and distance form the top of the head to the floor is measured in cm.
Anthropometric measurements: weight | Measurements will be made at baseline and after the intervention (3 months)
  Weight in Kg is measured usind a scale
Anthropometric measurements: perimeters | Measurements will be made at baseline and after the intervention (3 months)
  Hip and waist perimeters are measured (in cm) using a tape measure.
Frailty Tilburg | Measurements will be made at baseline and after the intervention (3 months)
  Tilburg Frailty index estimates frailty. Construct: Multidimensional frailty. Scale range (total score): 0-15 (the higher, the worse).
  References:
  Gobbens et al., 2010. The Tilburg Frailty Indicator: psychometric properties. J Am Med Dir Assoc. 11(5):344-55. doi:10.1016/j.jamda.2009.11.003.
Frailty Fried | Measurements will be made at baseline and after the intervention (3 months)
  Fried's Frailty index estimates frailty.
  Construct: Frailty phenotype. Scale range (total score): 0-5 (the higher, the worse).
  References:
  Fried et al., 2001. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 56(3):M146-56. doi: 10.1093/gerona/56.3.M146.
Falls | Measurements will be made at baseline and after the intervention (3 months)
  Number of falls will be recorded from the medical records. Record from the last year and during the intervention will be recorded
Deaths | From baseline, during the intervention (3 months)
  Number of deaths will be recorded during the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Susana M Gil, MD, PhD, Principal Investigator — University of the Basque Country (UPV/EHU)
Locations (1):
- Basque Country, Leioa, Bizkaia, Spain